CLINICAL TRIAL: NCT01044979
Title: Measurements of Colloid Osmotic Pressure in Interstitial Fluid and Plasma, a Methodological Study
Brief Title: Measurements of Colloid Osmotic Pressure in Interstitial Fluid and Plasma
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 071223
Record Dates: First submitted 2009-12-17; First posted 2010-01-08 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Colloid Osmotic Pressure
Keywords: Colloid osmotic pressure in interstitial fluid; Colloid osmotic pressure in plasma; Protein fractions in interstitial fluid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and interstitial fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate a method of sampling interstitial fluid from subcutaneous sewn wicks.

DETAILED DESCRIPTION:
Fluid loss from circulating plasma volume is one of the contributors of oedema formation. Measurement of colloid osmotic pressure (COP) both in plasma and in interstitial fluid can be utilised in planing of fluid therapy in patients with oedema. Different methods of sampling interstitial fluid are well validated in animal models, but not in human. Sampling of interstitial fluid by subcutaneous sewn wicks is a well-known method and can be painful. Local anaesthetics can reduce pain. By comparing interstitial fluid taken from areas with or without application of local anaesthetics, a possible influence in COP values can be detected.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years

Exclusion Criteria:

* Ongoing illness
* Medication

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers over 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Colloid osmotic pressure | 60 and 90 minuttes after implanting wicks

CONTACTS AND LOCATIONS:
Overall Officials: Hans Joergen T Guthe, MD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Bergen, Norway

REFERENCES:
- [Derived] Guthe HJ, Nedrebo T, Tenstad O, Wiig H, Berg A. Effect of topical anaesthetics on interstitial colloid osmotic pressure in human subcutaneous tissue sampled by wick technique. PLoS One. 2012;7(2):e31332. doi: 10.1371/journal.pone.0031332. Epub 2012 Feb 14. PMID 22348071